CLINICAL TRIAL: NCT04607655
Title: GULLIVER-1 - A Randomised, Double-Blind, Placebo Controlled, Phase Ib, 12-week Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Administered GB1211 in Participants With Suspected or Confirmed Non-alcoholic Steatohepatitis (NASH) and Liver Fibrosis
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Administered GB1211 in Participants With Suspected or Confirmed Non-alcoholic Steatohepatitis (NASH) and Liver Fibrosis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to COVID-19 pandemic and change in the clinical development strategy for the GB1211 compound
Sponsor: Galecto Biotech AB (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GULLIVER-1; 2020-000687-34 (EudraCT Number)
Record Dates: First submitted 2020-10-19; First posted 2020-10-29 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-10

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: GB1211; Non-alcoholic Steatohepatitis; NASH; Liver Fibrosis; Galectin-3 Inhibitor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: All subjects eligible for the study will be randomised into one of the three treatment arms:
  A. GB1211 100 mg twice a day B. GB1211 10 mg twice a day C. Placebo twice a day
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind study. The blinding will be maintained throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral GB1211, 100 mg, twice a day (Experimental): GB1211 is a galectin-3 inhibitor an orally available small molecule anti-fibrotic. It is administered orally twice a day.
  Interventions: Drug: GB1211
- Oral GB1211, 10 mg, twice a day (Experimental): GB1211 is a galectin-3 inhibitor an orally available small molecule anti-fibrotic. It is administered orally twice a day.
  Interventions: Drug: GB1211
- Oral GB1211, Placebo, twice a day (Placebo Comparator): Placebo is administered as inhalation once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB1211 — GB1211 is a galectin-3 inhibitor an orally available small molecule anti-fibrotic. It is administered orally twice a day.
  Arms: Oral GB1211, 10 mg, twice a day; Oral GB1211, 100 mg, twice a day
Drug: Placebo — Placebo is administered as inhalation once a day
  Arms: Oral GB1211, Placebo, twice a day

SUMMARY:
This study is a randomised, double-blind, placebo controlled, phase Ib trial in subjects with suspected or confirmed non-alcoholic steatohepatitis (NASH) and liver fibrosis

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of orally administered GB1211 a gelectin-3 inhibitor over 12 weeks. Participants will receive two doses of GB1211, each given twice per day and compared to placebo in participants with fibrotic NASH

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, ≥ 18 and ≤ 75 years of age at enrolment. 2. Body mass index (BMI) of ≥ 25.0 and ≤45.0 kg/m2 3. Diagnosis of suspected NASH and liver fibrosis (Chalasani et al. 2012):

a. Evidence of hepatic steatosis within the 24 weeks prior to Screening: i. magnetic resonance imaging (MRI PDFF) suggesting liver fat ≥ 8% or ii. ultrasound (US) indicating fatty liver or iii. FibroScan Controlled Attenuation Parameter (CAP) > 270 dB/m. iv. in participants without a documented history of fatty liver, a FibroScan CAP or US can be performed at Screening. Participants with FibroScan CAP > 270 dB/m or US indicating fatty liver are eligible AND b. Metabolic risk factors: i. Metabolic syndrome (Adult Treatment Panel III definition) requires three or more of the following five disorders (Grundy et al. 2005):

1. elevated waist circumference (≥102 cm in men and ≥88 cm in women),
2. hypertriglyceridemia (≥1.7 mmol/l),
3. low HDL cholesterol level (<1.03 mmol/l in men and <1.3 mmol/l in women),
4. high blood pressure (systolic blood pressure ≥130 mmHg and/or diastolic blood pressure ≥85 mmHg and/or pharmacological treatment)
5. elevated fasting glucose (≥5.6 mmol/l and/or pharmacological treatment) ii. OR T2DM (defined as stable diabetes with glycosylated haemoglobin [HbA1c] ≤ 9.5%) OR A diagnosis of confirmed NASH and liver fibrosis based on a biopsy within 12-months of Screening

4. Liver stiffness as measured by transient elastography (FibroScan) ≥ 8.5 KPa 5. Women of non-childbearing potential defined as permanently sterile (see Appendix 4) or postmenopausal (see Appendix 4) or Women considered to be of childbearing potential who agree to use highly effective birth control methods until 90 days after the Follow-up visit (see Appendix 4) 6. Males will agree to use contraception throughout the study and until 90-days after the Follow-up visit 7. Male participants must agree to refrain from sperm donation and females should refrain from ova donation from the date of Randomisation (Day -1) until 90 days after the Follow up visit 8. Able to comprehend and willing to sign an ICF and to abide by the study restrictions

Exclusion Criteria:

1. Any other causes for secondary hepatic fat accumulation such as significant alcohol consumption, use of steatogenic medication or hereditary disorders
2. The following clinical laboratory results at Screening:

   1. ALT > 200 U/L
   2. AST > 200 U/L
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair will be allowed)
4. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Randomisation
5. Positive hepatitis panel and/or positive HIV test
6. Evidence of acute Hepatitis A virus (HAV) and a positive serological test for anti-HAV IgM antibodies
7. Estimated glomerular filtration rate (eGFR) < 60 mL/[min*1.73 m²] at Screening
8. Use or intend to use slow release medications/products considered to still be active within 14 days prior to Randomisation, unless deemed acceptable by the Investigator (or Designee)
9. Participant taking any antidiabetic medications, with the exception of metformin and sulfonylureas within 3 months prior to Screening
10. Have previously completed or withdrawn from this study investigating GB1211 and have previously received the investigational product
11. Participant who, in the opinion of the Investigator (or Designee), should not participate in this study
12. Vulnerable/institutionalised patients
13. Patients related to PI/site staff

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of GB1211 | 12 Weeks
  Incidence and severity of adverse events as reported by investigators
Safety and Tolerability of GB1211 | 12 Weeks
  Incidence of laboratory abnormalities as measured by haematology, clinical chemistry and urinalysis
Safety and Tolerability of GB1211 | 12 Weeks
  Physical examination abnormalities measured by vital signs and 12 lead ECG

SECONDARY OUTCOMES:
Pharmacokinetics of GB1211 | 12 Weeks
  AUC over a dosing interval (AUC0-τ)
Pharmacokinetics of GB1211 | 12 Weeks
  Cmax
Pharmacokinetics of GB1211 | 12 Weeks
  Tmax
Pharmacokinetics of GB1211 | 12 Weeks
  t1/2
Pharmacokinetics of GB1211 | 12 Weeks
  Minimum observed plasma concentration (Cmin)
Pharmacokinetics of GB1211 | 12 Weeks
  Observed accumulation ratio based on AUC0-τ (RAAUC0-τ)
Pharmacokinetics of GB1211 | 12 Weeks
  Observed accumulation ratio based on Cmax (RACmax)
Pharmacokinetics of GB1211 | 12 Weeks
  Volume of distribution and rate of elimination

CONTACTS AND LOCATIONS:
Overall Officials: Michael Charlton, MD, Principal Investigator — The University of Chicago Biological Sciences

IPD SHARING:
Plan to Share IPD: No